CLINICAL TRIAL: NCT06519097
Title: A Randomized, Placebo-Controlled Trial of Tocotrienol in the Prevention of Pancreatic Intraductal Papillary Mucinous Neoplasm Progression
Brief Title: Study of IPMN Progression Prevention With Tocotrienol (SIPP-T3)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American River Nutrition, LLC (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCC-21791; R01CA263575 (NIH)
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Neoplasm of Pancreas; IPMN, Pancreatic
Keywords: Papillary Mucinous Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Intraductal Neoplasms | interventions — tocotrienol, delta

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: All eligible patients will be allocated randomly to one of 2 groups, the DT3 group and the Placebo group. Surgeons, medical oncologists, advanced practice professionals (APPs) (nurse practitioners and physician assistants) at the follow-up outpatient clinics, and patients will be blinded to the allocation. Patients in the DT3 group shall receive oral DT3 400 mg twice per day, and those in the placebo group shall receive oral placebo twice per day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin E Delta-tocotrienol (DT3) (Experimental): Patients will be given DT3 orally (by mouth) twice daily for 3 years
  Interventions: Drug: Vitamin E Delta Tocotrienol
- Placebo (Active Comparator): Patients will be given a placebo (a substance that looks like the study drug, but contains not active ingredients) orally (by mouth) twice daily for 3 years
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin E Delta Tocotrienol — Tocotrienols are natural vitamin E compounds that are known to have a neuroprotective effect at nanomolar concentration and anti-carcinogenic effect at micromolar concentration.
  400 mg orally, twice daily
  Other Names: DT3
  Arms: Vitamin E Delta-tocotrienol (DT3)
Other: Placebo — Placebo contains no active ingredients.
  465 mg pure olive oil orally, twice daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial, investigating whether treatment with δ-tocotrienol (a.k.a. Delta-tocotrienol, abbreviated as DT3) will prevent the progression of Intraductal Papillary Mucinous Neoplasm (IPMN) of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age ≥18 years.
* Evidence of IPMN as confirmed by MRI/Magnetic Resonance Cholangiopancreatography (MRCP) or pathology with biomarker results from Endoscopic Ultrasound-Guided Fine Needle Aspiration (EUS/FNA).
* IPMN must be suitable for active surveillance as defined by the international Kyoto guidelines and the European guidelines. Patients eligible for our study will have IPMN with no "high-risk stigmata" and no "worrisome features" and also have a neoplasm size of 1-<3 cm.
* Able to complete all of the periodic activities of active surveillance as defined by the international Kyoto guidelines (2024) (Appendix VII) and the European guidelines (clinic visit evaluation, blood work, MRI/MRCP, and EUS).
* Eastern Cooperative Oncology Group = 0-2.
* Participants must have adequate organ and marrow function.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should undergo a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification (see Appendix VI). To be eligible for this trial, participants should be class I-II.
* Agrees to avoid dietary sources of increased DT3 and abstain from consuming non-study DT3 supplements, any other dietary supplements, herbal remedies and over the counter (OTC) medicines (except use of aspirin for which data will be collected in Oncore) beginning 3 days prior to start of study drug and throughout duration of the study. DT3 levels are extremely low in normal foods. Therefore, no specific foods need to be avoided. All supportive care medications, e.g., antiemetics, antidiarrheals growth factors etc. may be used at the discretion of the treating physician and according to institutional guidelines.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must agree to refrain from getting pregnant, breastfeeding or fathering a child for the duration of the study. Female participants of child-bearing potential and male participants with a female partner of child-bearing potential must agree to use an effective birth control method, as specified in the informed consent form, throughout the study and for 6 months following the last dose of DT3. For purposes of this study, child-bearing potential is defined as a premenopausal woman without permanent sterilization who has the potential to become pregnant by being exposed to sexual intercourse with a non-sterilized male partner. Examples of birth control methods include:

  * Oral birth control pills
  * Birth control patch
  * Implanted (injectable contraceptive hormones or mechanical products such as intrauterine device)
  * Barrier methods (such as: diaphragm, condoms, or spermicides)
  * Tubal ligation or vasectomy
  * Abstinence (no sexual intercourse)

Exclusion Criteria:

* Evidence of Pancreatic Ductal Adenocarcinoma (PDAO or other cancers (excluding non-melanoma skin cancer) or metastatic disease.
* Concurrent systemic chemotherapy for any other cancer.
* Use of increased dietary sources of DT3, non-study DT3 supplements, any other dietary supplements, herbal remedies and OTC medicines (except use of aspirin for which data will be collected in Oncore) which may affect the study outcome unless the participant is willing to discontinue taking them 3 days prior to start of study drug DT3 and for the duration of the study. DT3 levels are extremely low in normal foods. Therefore, no specific foods need to be avoided.
* Participants may not be receiving any other investigational agents.
* History of allergic reaction attributed to vitamins.
* Patient is lactating, pregnant or planning to become pregnant during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
IPMN Progression Free Survival (iPFS) | Up to 60 Months
  IPMN progression free survival (iPFS) defined as duration from date of randomization to date of event (IPMN progression), pursuant to the international Kyoto guidelines and the European guidelines.
  IPMN will be considered as having progressed if any one or more of the following features occur:
  (i) increase in size of > 1 mm; (ii) development of any worrisome feature (growth rate ≥ 5 mm/ 2 years, main pancreatic duct dilatation from 5-9 mm, acute pancreatitis caused by IPMN, enhancing mural nodule < 5 mm, increased serum CA 19-9 ≥ 37 U/ml, and cyst diameter ≥ 3 cm); or development of any high-risk stigmata (positive cytology for malignancy, solid mass, tumor related jaundice, enhancing mural nodule ≥ 5 mm, and main pancreatic duct dilatation ≥ 10 mm).

SECONDARY OUTCOMES:
Time to Surgical Intervention (TSI) | Up to 36 Months
  The time to surgical intervention (TSI), defined as duration from date of randomization to date of event (Surgical Intervention for IPMN).
Bioavailability and Biodistribution | Baseline, Month 6, 12, 24 and 36
  The difference of DT3 and metabolite levels will be measured in IPMN cyst fluid, plasma, and urine before and after treatment in the DT3 arm.
  The analytes will be quantified by comparing the peak heights with those of the serum, urine, and cyst standards.
Acceptability of DT3 Treatment | Baseline, Month 6, 12, 24 and 36
  Quality of life (QoL) and functional health and well-being from the patient's point of view (SF-36v2) will be evaluated before the start of treatment and at each follow-up.
  DT3 acceptability will be analyzed as a change of SF36 score before and after treatment to assess quality of life.
  Overall compliance of 80% adherence to study agent intake will be required during the 3-year intervention.
Adherence of DT3 Treatment | Baseline, Month 6, 12, 24 and 36
  To determine the adherence of DT3 treatment, participants will be provided with the Study Agent Intake and Symptom Log that the subject will complete daily.
  Overall compliance of 80% adherence to study agent intake will be required during the 3-year intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mokenge P Malafa, MD, FACS, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/